CLINICAL TRIAL: NCT04234516
Title: Functional Brain Mechanisms Underlying the Anti-suicidal Effects of Buprenorphine in Opioid Use Disorder
Brief Title: Anti-suicidal Effects of Buprenorphine in Opioid Use Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI leaving the institute
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Mina.Rizk, Paul Janssen Postdoctoral Fellow, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB #7855
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Opioid-use Disorder; Suicidal Ideation
MeSH Terms: conditions — Opioid-Related Disorders; Suicidal Ideation | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind, double dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buprenorphine (Active Comparator): Sublingual buprenorphine-naloxone films
  Interventions: Drug: Buprenorphine/Naloxone 8/2 milligram (mg) Sublingual Film
- Morphine (Active Comparator): Oral morphine sulphate tablets
  Interventions: Drug: Morphine Sulfate 30 mg

INTERVENTIONS:
Drug: Buprenorphine/Naloxone 8/2 milligram (mg) Sublingual Film — 3 x 8 mg sublingual buprenorphine/naloxone films wrapped inside one Listerine strip at 8 pm daily + oral placebo pills q.i.d.
  Other Names: buprenorphine
  Arms: Buprenorphine
Drug: Morphine Sulfate 30 mg — oral morphine sulphate 30 mg immediate release tablets q.i.d. + two sublingual Listerine strips at 8 pm
  Other Names: morphine
  Arms: Morphine

SUMMARY:
The study aims to examine the effect of buprenorphine on suicidal ideation in individuals with opioid use disorder, and to investigate the functional brain activity related to its potential anti-suicidal effect.

DETAILED DESCRIPTION:
The current opioid epidemic is an urgent public health problem, contributing significantly to the climbing U.S. suicide rates over the past two decades.

Although initially rewarding, chronic opioid use leads to tolerance and escalating negative affective states. This may promote suicidal ideation and may further impair decision-making functions leading to suicidal behavior.

Buprenorphine, a treatment for opioid use disorder (OUD), has promise in reducing suicidal ideation. However, the neural mechanism of its anti-suicidal properties remains unknown. Blocking kappa opioid receptors is one mechanism of buprenorphine hypothesized to reverse the negative emotional sensitivity in OUD and thus may underlie its anti-suicidal effects.

In this morphine-controlled study, we will examine the effect of buprenorphine on the functional activity of brain regions involved in negative emotional reactivity and investigate whether this effect is associated with its anti-suicidal properties.

Buprenorphine has a different mechanism of action than currently available antidepressants and anti-suicidal medications. Understanding this mechanism can help refine its use in this context. Success will guide a future larger study to elucidate molecular mechanisms underlying anti-suicidal properties of buprenorphine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years old
* Current opioid use disorder (mild, moderate or severe)
* Seeking treatment for opioid use disorder and willing to accept agonist-based therapy and be stabilized on buprenorphine when study is over
* Active suicidal ideation
* Participant must agree to voluntary admission to New York State Psychiatric Institute (NYSPI) inpatient research unit with confirmed bed availability
* Capacity to provide informed consent

Exclusion Criteria:

* Presence of chronic pain of sufficient severity as to require ongoing pain management with opioids
* Current active psychosis or mania
* Current moderate-severe alcohol, benzodiazepine, or other drug use likely to require a medical detoxification
* Unstable epilepsy or other neurological disorder
* A history of prior head trauma with evidence of cognitive impairment. Participants who endorse a history of prior head trauma will be administered Trail-making A and B test. Those who score 1.5 standard deviations below the mean on Trail- making A or B will be excluded from study participation
* Active significant medical illness that, in the opinion of the study physician, would make study participation hazardous to the participant or compromise study findings or would prevent the participant from completing the study (e.g., uncompensated heart failure, cirrhosis or end-stage liver disease)
* Liver Function Tests (ALT, AST) greater than 5 times upper limit of normal
* On methadone-maintenance therapy
* Contraindication to any study treatment (e.g., Known allergy or sensitivity to buprenorphine)
* Pending legal action or other reasons that might prevent an individual from completing the study
* If female, currently pregnant or breastfeeding, or planning on conception
* Inadequate understanding of English
* Metal implants or paramagnetic objects contained within the body (including heart pacemaker, shrapnel, or surgical prostheses) which may present a risk to the subject or interfere with the MRI scan
* Claustrophobia significant enough to interfere with MRI scanning
* Weight over 350 lbs or inability to fit into MRI scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Changes in Beck Scale for Suicidal Ideation (SSI) scores from baseline to Week 2 post-treatment | 2 weeks
  Clinician-based questionnaire measuring level of suicidal ideas over the last 7 days; 21 items scored 0 to 2; total score ranges from 0 to 38 (last 2 items not counted), higher scores mean more intense suicidal ideas.
Changes in functional magnetic resonance imaging (fMRI) blood oxygen-level dependent (BOLD) signal in the amygdala in response to negative vs. neutral pictures from baseline to Week 2 post-treatment | 2 weeks
  fMRI negative picture task administered at baseline and week 2 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mina M Rizk, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No